CLINICAL TRIAL: NCT01456091
Title: Evaluation of the Efficacy of the AIM (Adult Identity Mentoring) 4 Teen Moms Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Children's Hospital Los Angeles (Other); ETR Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MPR06549-2
Record Dates: First submitted 2011-10-18; First posted 2011-10-20 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Pregnancy
Keywords: adolescent pregnancy; adolescent birth; rapid repeat pregnancy; rapid repeat birth; youth development; Pregnancy in Adolescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AIM 4 Teen Moms (Experimental)
  Interventions: Behavioral: AIM 4 Teen Moms
- Control (No Intervention)

INTERVENTIONS:
Behavioral: AIM 4 Teen Moms — The AIM (Adult Identity Mentoring) 4 Teen Moms program is a combination of individual and small group sessions intervention that encourages parenting young women ages 15-19 years old to delay rapid repeat pregnancies for 24 months or later.
  Arms: AIM 4 Teen Moms

SUMMARY:
The purpose of this study is to evaluate the efficacy of the AIM 4 Teen Moms program in increasing the use of long-term contraceptives, in improving adherence to contraceptives and in preventing rapid repeat pregnancies among parenting adolescents.

DETAILED DESCRIPTION:
This study uses a randomized controlled design to evaluate the efficacy of AIM (Adult Identity Mentoring) 4 Teen Moms in reducing the incidence of rapid repeat pregnancies and associated sexual risk behavior. The AIM 4 Teen Moms program is a combination of individual and small group sessions intervention that encourages parenting young women ages 15-19 years old to delay rapid repeat pregnancies for 24 months or later. It consists of seven individual 1-hour long sessions (generally conducted in the participant's home) and two 90-minute group sessions delivered over a 12 week period. Study participants will be adolescent mothers receiving services from California's Adolescent Family Life or Cal-Learn programs in the Los Angeles County area. There will be no intervention delivered to members of the control group. This study is being conducted as part of the national Evaluation of Adolescent Pregnancy Prevention Approaches funded by the U.S. Department of Health and Human Services' Office of Adolescent Health.

ELIGIBILITY:
Inclusion Criteria:

* Beneficiaries of California's Adolescent Family Life or Cal-Learn programs in the Los Angeles County area
* Female
* 15 - 19 years old
* Has a child between the ages 1 and 6 months at program start
* English or Spanish speaker

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 954 (Actual)
Dates: Start 2011-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Incidence of repeat pregnancy | 24 months after baseline

SECONDARY OUTCOMES:
Adherence to contraception | 12 months after baseline
Adherence to contraception | 24 months after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Trenholm, Ph.D., Principal Investigator — Mathematica Policy Research; Reginald Covington, Ph.D., Principal Investigator — Mathematica Policy Research; Pamela Drake, Ph.D., Principal Investigator — ETR Associates
Locations (4):
- United States (4):
  - El Nido Family Centers-Manchester, Los Angeles, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - El Nido Family Centers-Mission Hills, Mission Hills, California
  - El Nido Family Centers-Pacoima, Pacoima, California

REFERENCES:
- [Derived] Cederbaum JA, Yoon Y, Lee JO, Desai M, Brown K, Clark L. AIM for Teen Moms: Social Support's Role in Contraception Use Among Young Mothers. J Adolesc Health. 2022 Jul;71(1):78-85. doi: 10.1016/j.jadohealth.2022.01.225. Epub 2022 Mar 15. PMID 35300930